CLINICAL TRIAL: NCT06787053
Title: Selecting Hypoxic Tumours for Treatment Modification
Acronym: SELECT
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Ananya Choudhury, Professor, University of Manchester
Other Study IDs: 24_DOG13_38
Record Dates: First submitted 2024-12-13; First posted 2025-01-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-01

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; Prostate Cancer
Keywords: Hypoxia; Bladder; Cervix; Prostate; Hypoxia Modification
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and formalin-fixed paraffin-embedded (FFPE) tumour biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Bladder: Patients diagnosed with bladder cancer
- Prostate: Patients diagnosed with prostate cancer
- Cervix: Patients diagnosed with cervical cancer

SUMMARY:
Approximately 50% of cancer patients with solid tumours will be treated with radiotherapy. A significant proportion (>25%) of patients have hypoxic tumours which respond poorly to radiotherapy. Hypoxic tumours have a poor prognosis. This can be improved with treatment intensification. Treatment intensification can be modification with CON (breathing O2-enriched air + oral administration of nicotinamide), chemoradiosensitisation, radiation dose-escalation or additional systemic treatments, significantly improving response of the tumours to radiotherapy. However, there are currently no clinically approved biomarkers to identify hypoxic tumours. Our group has developed and validated gene-expression signature-based biomarkers that identify patients with hypoxic bladder, head and neck , prostate, sarcoma and lung cancers. The bladder cancer gene-expression hypoxia signature has been shown to predict benefit from hypoxia modification using RNA from archived tumour tissue. The main purpose of this study is to demonstrate in at least two cancer types that the hypoxia biomarker predicts benefit from hypoxia modification in real-time.

DETAILED DESCRIPTION:
Research Question: Can hypoxia biomarkers personalised treatment improve cancer outcomes?

Cancers that are hypoxic (have a high percentage of regions of low local O2 concentration) are refractory to radiotherapy but benefit from hypoxia modification. However, there are no biomarkers to identify patients with hypoxic tumours. The gold standard for determining tissue O2 concentration is the O2-electrode which takes measurements at several sites within the tumour. However, this necessitates insertion of a needle into multiple regions of the tumour so is invasive and provides only a localised hypoxia status. Other hypoxia biomarkers that identify hypoxia have been derived from cell surface protein expression, gene expression or imaging outputs. Proteins expressed on the tumour cell surface of hypoxic cells include CA9 and glut1 but the expression of these proteins is not specific to hypoxia and is highly heterogeneous within tumours. Whilst expression of HIF1 by hypoxic tumours has been shown not to predict benefit from hypoxia-modification. Gene signatures are a set of genes in which the collective changed expression has been validated to demonstrate diagnosis, prognosis or predict therapeutic response. Gene expression is consistently altered across tumours with high hypoxic fractions meaning that they are robust indicators of hypoxia status.

Using RNA extracted from archived material (Formalin fixed paraffin embedded tumour tissue) our gene-expression signature-based biomarkers for bladder, head and neck, prostate, sarcoma, cervical and lung cancers have been validated by demonstrated prognosis in each of the cancer groups. Further the 24 gene bladder cancer hypoxia signature has been shown to be predictive of benefit from hypoxia modification for patients with hypoxic tumours receiving radiotherapy. A recent review of predictive biomarkers in cancer treatment has shown that this is the only predictive biomarker for hypoxia-modification during radiotherapy.

Hypoxic regions in tumours can also be identified using MRI techniques including O2-senstive MRI (OE-MRI) and Intravoxel incoherent motion imaging. Combining imaging with gene expression data results in more accurate assessment of hypoxic status and identify tumour subtype which further contributes to personalised clinical decisions. MRI-based techniques also facilitate localized personalization approaches, e.g., for hypoxia-directed focal radiotherapy dose escalation.

Primary Question/Objective:

Short objective; to establish trials to test if personalised use of established hypoxia-targeted treatments with radiotherapy improves survival and work with the North West Genomics Hub to progress implementing our tissue hypoxia test for delivery across the NHS.

Medium objective; integrate MR imaging in the workflow for measuring hypoxia in at least two tumour sites.

Secondary Question/Objective:

* Integrate radiological parameters with the hypoxia biomarker for personalising treatment.
* Can blood-based biomarkers be early response biomarkers.

ELIGIBILITY:
Inclusion Criteria:

This will be tumour site dependent.

Bladder:

* Older than age 18 years.
* Patients having radiotherapy at the Christie NHS Foundation Trust suitable for imaging on an MRI scanner.
* Able to give informed consent.

Cervix:

* Older than age 18 years.
* Patients having radiotherapy at the Christie NHS Foundation Trust suitable for imaging on an MRI scanner.
* Able to give informed consent.

Prostate:

* Older than age 18 years.
* Patients having radiotherapy at the Christie NHS Foundation Trust suitable for imaging on an MRI scanner.
* Able to give informed consent.

Exclusion Criteria:

This will be tumour site dependent

Bladder:

* Any contraindications to MRI identified after MRI safety screening including completion of an MRI Safety Screening Form.
* Unable to tolerate MRI scans.
* Pregnancy.

Cervix:

* Any contraindications to MRI identified after MRI safety screening including completion of an MRI Safety Screening Form.
* Unable to tolerate MRI scans.
* Pregnancy.

Prostate:

* Any contraindications to MRI identified after MRI safety screening including completion of an MRI Safety Screening Form.
* Unable to tolerate MRI scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient recruitment will be via the disease site clinics .
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Primary | Through to study completion, until May 2028
  To have collected the FFPE tumour blocks and generate the gene signature.

SECONDARY OUTCOMES:
Secondary Outcome Measure | end of the study in May 2028
  To have collected a total of at least 4 different patient blood samples which have corresponding MRI scans from each participant in this study undergoing imaging or treatment.
  To have developed and optimised MR sequences, which can be used across Manchester and Lancashire in at least two tumour sites.

CONTACTS AND LOCATIONS:
Overall Officials: Ananya Choudhury, Professor, Principal Investigator — University of Manchester
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Swartz JE, Smits HJG, Philippens MEP, de Bree R, H A M Kaanders J, Willems SM. Correlation and colocalization of HIF-1alpha and pimonidazole staining for hypoxia in laryngeal squamous cell carcinomas: A digital, single-cell-based analysis. Oral Oncol. 2022 May;128:105862. doi: 10.1016/j.oraloncology.2022.105862. Epub 2022 Apr 18. PMID 35447566
- [Background] Batis N, Brooks JM, Payne K, Sharma N, Nankivell P, Mehanna H. Lack of predictive tools for conventional and targeted cancer therapy: Barriers to biomarker development and clinical translation. Adv Drug Deliv Rev. 2021 Sep;176:113854. doi: 10.1016/j.addr.2021.113854. Epub 2021 Jun 27. PMID 34192550
- [Background] Yang L, Taylor J, Eustace A, Irlam JJ, Denley H, Hoskin PJ, Alsner J, Buffa FM, Harris AL, Choudhury A, West CML. A Gene Signature for Selecting Benefit from Hypoxia Modification of Radiotherapy for High-Risk Bladder Cancer Patients. Clin Cancer Res. 2017 Aug 15;23(16):4761-4768. doi: 10.1158/1078-0432.CCR-17-0038. Epub 2017 Apr 11. PMID 28400426
- [Background] Yang L, Roberts D, Takhar M, Erho N, Bibby BAS, Thiruthaneeswaran N, Bhandari V, Cheng WC, Haider S, McCorry AMB, McArt D, Jain S, Alshalalfa M, Ross A, Schaffer E, Den RB, Jeffrey Karnes R, Klein E, Hoskin PJ, Freedland SJ, Lamb AD, Neal DE, Buffa FM, Bristow RG, Boutros PC, Davicioni E, Choudhury A, West CML. Development and Validation of a 28-gene Hypoxia-related Prognostic Signature for Localized Prostate Cancer. EBioMedicine. 2018 May;31:182-189. doi: 10.1016/j.ebiom.2018.04.019. Epub 2018 Apr 23. PMID 29729848
- [Background] Lane B, Khan MT, Choudhury A, Salem A, West CML. Development and validation of a hypoxia-associated signature for lung adenocarcinoma. Sci Rep. 2022 Jan 25;12(1):1290. doi: 10.1038/s41598-022-05385-7. PMID 35079065
- [Background] Forker LJ, Bibby B, Yang L, Lane B, Irlam J, Mistry H, Khan M, Valentine H, Wylie J, Shenjere P, Leahy M, Gaunt P, Billingham L, Seddon BM, Grimer R, Robinson M, Choudhury A, West C. Technical development and validation of a clinically applicable microenvironment classifier as a biomarker of tumour hypoxia for soft tissue sarcoma. Br J Cancer. 2023 Jun;128(12):2307-2317. doi: 10.1038/s41416-023-02265-3. Epub 2023 Apr 21. PMID 37085598
- [Background] Eustace A, Mani N, Span PN, Irlam JJ, Taylor J, Betts GN, Denley H, Miller CJ, Homer JJ, Rojas AM, Hoskin PJ, Buffa FM, Harris AL, Kaanders JH, West CM. A 26-gene hypoxia signature predicts benefit from hypoxia-modifying therapy in laryngeal cancer but not bladder cancer. Clin Cancer Res. 2013 Sep 1;19(17):4879-88. doi: 10.1158/1078-0432.CCR-13-0542. Epub 2013 Jul 2. PMID 23820108